CLINICAL TRIAL: NCT01116102
Title: The INcreased Flow Utilizing Subcutaneously-Enabled Fluids Administration Technique 1A Study (INFUSE-AT 1A): A Randomized, Parallel Group Study to Evaluate the In-line Pressure, Flow Rate, Safety and Tolerability of Hylenex-facilitated Subcutaneous Fluid Administration In Healthy Volunteers Using Various Subcutaneous Infusion Techniques
Brief Title: Study of In-line Pressure Using Various Techniques of Subcutaneous Administration of Fluids Enabled by Human Recombinant Hyaluronidase (INFUSE-AT1A)
Acronym: INFUSE-AT1A
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Strategic business decision (not related to safety or efficacy concerns)
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1838-009
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Results first posted 2011-10-18 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Dehydration
Keywords: dehydration; fluid therapy; hyaluronoglucosaminidase; hyaluronidase; hypodermoclysis; clysis; subcutaneous hydration; subcutaneous rehydration; hyaluronan; rHuPH20
MeSH Terms: conditions — Dehydration | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 24 ga catheter, dose flush, single-step rate scheme (Experimental): Single 150 U subcutaneous (SC) dose of HYLENEX and 3 mL Lactated Ringer's solution flush administered through 24 gauge plastic catheter; followed by SC infusion of 1000 mL Lactated Ringer's solution via large-volume infusion pump at 250 mL/h for the first hour and 200 mL/hr for the remainder of the infusion.
  Interventions: Drug: Subcutaneous HYLENEX (recombinant human hyaluronidase) and Lactated Ringer's solution
- 24 ga catheter, no dose flush, single-step rate scheme (Experimental): Single 150 U subcutaneous (SC) dose of HYLENEX (without a Lactated Ringer's solution flush) administered through 24 gauge plastic catheter; followed by SC infusion of 1000 mL Lactated Ringer's solution via large-volume infusion pump at 250 mL/h for the first hour and 200 mL/hr for the remainder of the infusion.
  Interventions: Drug: Subcutaneous HYLENEX (recombinant human hyaluronidase) and Lactated Ringer's solution
- 24 ga catheter, dose flush, up-titrated rate scheme (Experimental): Single 150 U subcutaneous (SC) dose of HYLENEX and 3 mL Lactated Ringer's solution flush administered through 24 gauge plastic catheter; followed by SC infusion of 1000 mL Lactated Ringer's solution via large-volume infusion pump at 50 mL/h for the first 5 min, 100 mL/h for the next 5 min, 285 mL/h for the next 50 min and 200 mL/h for the remainder of the infusion.
  Interventions: Drug: Subcutaneous HYLENEX (recombinant human hyaluronidase) and Lactated Ringer's solution
- 24 ga catheter, no dose flush, up-titrated rate scheme (Experimental): Single 150 U subcutaneous (SC) dose of HYLENEX (without a Lactated Ringer's solution flush) administered through 24 gauge plastic catheter; followed by SC infusion of 1000 mL Lactated Ringer's solution via large-volume infusion pump at 50 mL/h for the first 5 min, 100 mL/h for the next 5 min, 285 mL/h for the next 50 min and 200 mL/h for the remainder of the infusion.
  Interventions: Drug: Subcutaneous HYLENEX (recombinant human hyaluronidase) and Lactated Ringer's solution
- 25 ga needle, dose flush, single-step rate scheme (Experimental): Single 150 U subcutaneous (SC) dose of HYLENEX and 3 mL Lactated Ringer's solution flush administered through 25 gauge metal butterfly needle; followed by SC infusion of 1000 mL Lactated Ringer's solution via large-volume infusion pump at 250 mL/h for the first hour and 200 mL/hr for the remainder of the infusion.
  Interventions: Drug: Subcutaneous HYLENEX (recombinant human hyaluronidase) and Lactated Ringer's solution
- 25 ga needle, no dose flush, single-step rate scheme (Experimental): Single 150 U subcutaneous (SC) dose of HYLENEX (without a Lactated Ringer's solution flush) administered through 25 gauge metal butterfly needle; followed by SC infusion of 1000 mL Lactated Ringer's solution via large-volume infusion pump at 250 mL/h for the first hour and 200 mL/hr for the remainder of the infusion.
  Interventions: Drug: Subcutaneous HYLENEX (recombinant human hyaluronidase) and Lactated Ringer's solution
- 25 ga needle, dose flush, up-titrated rate scheme (Experimental): Single 150 U subcutaneous (SC) dose of HYLENEX and 3 mL Lactated Ringer's solution flush administered through 25 gauge metal butterfly needle; followed by SC infusion of 1000 mL Lactated Ringer's solution via large-volume infusion pump at 50 mL/h for the first 5 min, 100 mL/h for the next 5 min, 285 mL/h for the next 50 min and 200 mL/h for the remainder of the infusion.
  Interventions: Drug: Subcutaneous HYLENEX (recombinant human hyaluronidase) and Lactated Ringer's solution
- 25 ga needle, no dose flush, up-titrated rate scheme (Experimental): Single 150 U subcutaneous (SC) dose of HYLENEX (without a Lactated Ringer's solution flush) administered through 25 gauge metal butterfly needle; followed by SC infusion of 1000 mL Lactated Ringer's solution via large-volume infusion pump at 50 mL/h for the first 5 min, 100 mL/h for the next 5 min, 285 mL/h for the next 50 min and 200 mL/h for the remainder of the infusion.
  Interventions: Drug: Subcutaneous HYLENEX (recombinant human hyaluronidase) and Lactated Ringer's solution

INTERVENTIONS:
Drug: Subcutaneous HYLENEX (recombinant human hyaluronidase) and Lactated Ringer's solution — Subcutaneous administration of 150 U HYLENEX, followed by 1000 mL Lactated Ringer's solution
  Other Names: rHuPH20; LR solution

SUMMARY:
The purpose is to characterize the in-line pressure profiles associated with several infusion technique factors during subcutaneous (SC) infusion of Lactated Ringer's solution, preceded by recombinant human hyaluronidase (hylenex). The safety and tolerability of hylenex-augmented SC infusion of Lactated Ringer's solution fluid is also being evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 60 years, inclusive.
* Body mass index 19.0 to 35.0 kg/m2
* Intact normal skin without potentially obscuring tattoos, pigmentation, or lesions on the upper back in the area intended for infusion
* Free from any clinically significant abnormality on the basis of medical/medication history or physical examination
* Vital signs and clinical laboratory parameters within normal range or, if outside normal range, deemed not clinically significant
* Negative urine drug and alcohol screens.

Exclusion Criteria:

* Upper back pathology that could interfere with study outcome.
* History of congestive heart failure, known coronary heart disease, active or recent pulmonary disease, or renal insufficiency.
* Rales on lung auscultation.
* Known allergy to hyaluronidase or any other ingredient in the formulation of hylenex recombinant
* Treatment with furosemide, benzodiazepines, or phenytoin.
* Pregnancy or breastfeeding.
* Exposure to any experimental drug within 30 days prior to study admission, or previous participation in this study.
* Any other reason which, in the investigator's opinion, would prevent the safe participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Harb, MD, MPH, Study Director — Baxter Healthcare Corporation
Locations (1):
- Kendle International, Inc. Drug Study Unit, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 24 ga Catheter, Dose Flush, Single-step Rate Scheme | 24 ga Catheter, No Dose Flush, Single-step Rate Scheme | 24 ga Catheter, Dose Flush, Up-titrated Rate Scheme | 24 ga Catheter, No Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, Dose Flush, Single-step Rate Scheme | 25 ga Needle, No Dose Flush, Single-step Rate Scheme | 25 ga Needle, Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, No Dose Flush, Up-titrated Rate Scheme
Started | 2 | 3 | 3 | 3 | 2 | 2 | 2 | 3
Completed | 2 | 3 | 3 | 3 | 2 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24 ga Catheter, Dose Flush, Single-step Rate Scheme | 24 ga Catheter, No Dose Flush, Single-step Rate Scheme | 24 ga Catheter, Dose Flush, Up-titrated Rate Scheme | 24 ga Catheter, No Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, Dose Flush, Single-step Rate Scheme | 25 ga Needle, No Dose Flush, Single-step Rate Scheme | 25 ga Needle, Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, No Dose Flush, Up-titrated Rate Scheme | Total
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 2 | 2 | 2 | 3 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 3 | 3 | 2 | 2 | 2 | 3 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Full Range); unit: years] | 45.9 [33.5 to 58.3] | 32.6 [25.4 to 36.7] | 39.6 [21.4 to 50.0] | 29.3 [19.9 to 46.4] | 35.4 [20.3 to 50.5] | 39.7 [37.0 to 42.4] | 28.2 [24.1 to 32.3] | 20.9 [19.9 to 21.9] | 33.3 [19.9 to 58.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 0 | 12
  Male | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 3 | 3 | 2 | 2 | 2 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured In-line Fluid Pressure
Description: Maximum fluid pressure measured (15 sec period) in delivery line during subcutaneous fluid infusion at specified time point after start of infusion
Time Frame: each minute for the first 15 minutes of fluid infusion, every 5 minutes for the next 45 minutes of infusion, and every 15 minutes thereafter until the end of infusion
Population: Per protocol (two subjects excluded due to technical error in in-line fluid pressure measurement)
Measure: Mean (Full Range); unit: psi
Arm/Group | 24 ga Catheter, Dose Flush, Single-step Rate Scheme | 24 ga Catheter, No Dose Flush, Single-step Rate Scheme | 24 ga Catheter, Dose Flush, Up-titrated Rate Scheme | 24 ga Catheter, No Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, Dose Flush, Single-step Rate Scheme | 25 ga Needle, No Dose Flush, Single-step Rate Scheme | 25 ga Needle, Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, No Dose Flush, Up-titrated Rate Scheme
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 1 | 2 | 3
psi
  1 min | 6.9 [2.6 to 11.1] | 3.0 [2.6 to 3.5] | 6.8 [3.1 to 10.6] | 5.0 [1.5 to 11.7] | 3.8 [3.7 to 3.8] | 2.8 [2.8 to 2.8] | 1.1 [1.0 to 1.2] | 3.0 [1.5 to 5.1]
  2 min | 6.8 [2.8 to 10.8] | 2.4 [2.1 to 2.7] | 7.8 [3.3 to 12.3] | 5.9 [1.0 to 14.2] | 4.1 [3.8 to 4.4] | 3.1 [3.1 to 3.1] | 1.1 [0.9 to 1.4] | 2.4 [1.1 to 4.7]
  3 min | 6.7 [2.8 to 10.6] | 2.1 [1.9 to 2.5] | 7.4 [3.5 to 11.2] | 6.1 [1.3 to 14.9] | 4.2 [4.1 to 4.4] | 3.2 [3.2 to 3.2] | 1.2 [1.1 to 1.3] | 2.5 [1.0 to 4.9]
  4 min | 6.6 [2.8 to 10.4] | 2.1 [1.8 to 2.5] | 7.3 [3.7 to 11.0] | 6.0 [1.0 to 15.9] | 4.3 [4.3 to 4.3] | 3.2 [3.2 to 3.2] | 1.0 [1.0 to 1.1] | 2.8 [1.6 to 4.7]
  5 min | 6.1 [2.7 to 9.5] | 2.6 [1.8 to 4.1] | 9.1 [7.7 to 10.6] | 5.7 [1.0 to 15.1] | 4.4 [4.3 to 4.4] | 3.2 [3.2 to 3.2] | 1.1 [1.1 to 1.1] | 2.5 [1.1 to 4.9]
  6 min | 6.2 [2.8 to 9.6] | 3.3 [1.8 to 6.0] | 8.0 [4.9 to 11.1] | 7.1 [1.4 to 18.4] | 4.1 [4.0 to 4.2] | 3.2 [3.2 to 3.2] | 2.2 [2.1 to 2.2] | 2.4 [2.2 to 2.5]
  7 min | 6.2 [2.8 to 9.7] | 3.2 [1.9 to 5.7] | 8.8 [3.4 to 14.1] | 7.1 [1.6 to 17.8] | 4.1 [4.1 to 4.2] | 3.2 [3.2 to 3.2] | 2.1 [2.1 to 2.2] | 3.8 [2.2 to 6.9]
  8 min | 6.4 [2.8 to 10.1] | 3.6 [2.0 to 5.9] | 9.0 [3.7 to 14.4] | 7.3 [2.8 to 16.1] | 4.2 [4.1 to 4.3] | 3.2 [3.2 to 3.2] | 2.1 [2.1 to 2.2] | 4.6 [2.1 to 7.6]
  9 min | 6.5 [2.8 to 10.2] | 3.8 [2.0 to 6.8] | 8.2 [2.9 to 13.5] | 7.0 [2.5 to 14.5] | 4.2 [4.2 to 4.2] | 3.2 [3.2 to 3.2] | 2.2 [2.1 to 2.3] | 4.1 [2.1 to 7.9]
  10 min | 6.5 [2.8 to 10.2] | 3.9 [1.9 to 6.7] | 7.7 [2.9 to 12.5] | 6.2 [2.4 to 12.6] | 4.1 [4.1 to 4.2] | 3.2 [3.2 to 3.2] | 2.2 [2.1 to 2.3] | 3.9 [2.1 to 7.4]
  11 min | 6.5 [2.7 to 10.3] | 3.7 [2.0 to 6.5] | 11.9 [5.5 to 18.2] | 7.6 [2.7 to 14.5] | 4.1 [4.0 to 4.2] | 3.2 [3.2 to 3.2] | 4.0 [3.9 to 4.0] | 6.4 [2.1 to 12.8]
  12 min | 6.7 [2.7 to 10.6] | 4.2 [1.6 to 8.9] | 13.6 [4.3 to 22.9] | 10.3 [2.2 to 21.2] | 4.1 [4.1 to 4.2] | 3.2 [3.2 to 3.2] | 3.8 [3.7 to 3.9] | 7.4 [2.1 to 13.0]
  13 min | 6.7 [2.7 to 10.7] | 3.6 [1.7 to 7.2] | 7.7 [3.1 to 12.2] | 10.5 [2.3 to 18.8] | 4.1 [4.0 to 4.2] | 3.2 [3.2 to 3.2] | 3.9 [3.8 to 4.0] | 7.0 [3.8 to 12.8]
  14 min | 6.6 [2.7 to 10.5] | 3.0 [1.7 to 5.2] | 3.5 [2.6 to 4.4] | 17.7 [2.1 to 34.2] | 4.1 [4.0 to 4.2] | 3.3 [3.3 to 3.3] | 3.6 [3.4 to 3.9] | 6.9 [3.8 to 11.4]
  15 min | 7.3 [3.5 to 11.0] | 4.0 [2.0 to 5.8] | 3.4 [2.6 to 4.2] | 15.8 [2.1 to 34.1] | 4.1 [4.1 to 4.2] | 3.2 [3.2 to 3.2] | 3.7 [3.5 to 3.9] | 6.5 [3.8 to 11.8]
  20 min | 7.3 [3.1 to 11.5] | 2.2 [1.7 to 3.0] | 3.3 [2.7 to 3.9] | 11.9 [1.8 to 26.3] | 4.1 [4.0 to 4.3] | 3.2 [3.2 to 3.2] | 3.6 [3.5 to 3.7] | 6.2 [3.8 to 10.9]
  25 min | 6.8 [3.1 to 10.4] | 2.4 [2.2 to 2.9] | 3.0 [2.0 to 4.1] | 8.7 [1.7 to 21.3] | 4.8 [4.3 to 5.4] | 3.2 [3.2 to 3.2] | 3.7 [3.7 to 3.8] | 6.1 [3.6 to 10.1]
  30 min | 5.8 [3.3 to 8.3] | 2.2 [1.8 to 2.8] | 8.4 [2.1 to 14.8] | 8.6 [1.7 to 21.2] | 4.8 [4.8 to 4.9] | 3.2 [3.2 to 3.2] | 3.8 [3.5 to 4.0] | 5.8 [3.6 to 9.8]
  35 min | 6.5 [3.3 to 9.8] | 2.7 [1.8 to 4.0] | 2.9 [2.0 to 3.9] | 10.9 [2.3 to 19.5] | 4.5 [4.5 to 4.5] | 3.3 [3.3 to 3.3] | 4.2 [3.4 to 5.1] | 6.4 [3.6 to 12.0]
  40 min | 7.0 [3.2 to 10.9] | 2.2 [2.1 to 2.3] | 2.9 [2.0 to 3.8] | 11.5 [2.1 to 20.8] | 4.6 [4.5 to 4.6] | 3.2 [3.2 to 3.2] | 3.4 [3.4 to 3.4] | 5.9 [3.6 to 10.6]
  45 min | 6.6 [2.8 to 10.4] | 2.3 [2.0 to 2.6] | 2.9 [2.0 to 3.9] | 7.4 [1.7 to 18.6] | 4.3 [4.1 to 4.6] | 3.2 [3.2 to 3.2] | 3.4 [3.3 to 3.5] | 5.8 [3.6 to 10.0]
  50 min | 6.4 [2.7 to 10.0] | 2.2 [1.8 to 2.6] | 3.0 [1.9 to 4.1] | 7.8 [1.6 to 19.8] | 4.5 [4.5 to 4.5] | 3.3 [3.3 to 3.3] | 3.4 [3.3 to 3.5] | 5.8 [3.5 to 10.1]
  55 min | 5.3 [2.8 to 7.9] | 2.4 [2.2 to 2.6] | 2.9 [1.9 to 3.8] | 7.9 [2.1 to 19.0] | 4.4 [4.3 to 4.5] | 3.2 [3.2 to 3.2] | 3.4 [3.2 to 3.5] | 6.0 [3.5 to 10.9]
  60 min | 5.3 [2.9 to 7.7] | 3.1 [1.9 to 4.3] | 2.9 [2.0 to 3.8] | 7.7 [1.5 to 19.3] | 3.7 [3.6 to 3.8] | 3.2 [3.2 to 3.2] | 3.4 [3.3 to 3.4] | 6.5 [3.5 to 12.2]
  75 min | 4.6 [2.6 to 6.7] | 2.6 [2.3 to 3.2] | 2.3 [1.8 to 2.8] | 5.9 [1.5 to 14.2] | 3.6 [3.0 to 4.1] | 2.8 [2.8 to 2.8] | 2.6 [2.6 to 2.7] | 7.8 [2.8 to 16.1]
  90 min | 4.1 [2.9 to 5.3] | 3.6 [2.4 to 4.5] | 2.1 [1.6 to 2.7] | 4.0 [1.3 to 8.9] | 3.5 [3.0 to 4.0] | 2.7 [2.7 to 2.7] | 2.7 [2.6 to 2.8] | 7.5 [2.7 to 16.7]
  105 min | 5.0 [2.9 to 7.1] | 2.7 [2.1 to 3.2] | 2.2 [1.7 to 2.7] | 4.5 [1.2 to 10.5] | 4.0 [3.1 to 4.9] | 2.7 [2.7 to 2.7] | 2.6 [2.6 to 2.6] | 6.3 [2.7 to 13.0]
  120 min | 3.4 [2.7 to 4.1] | 2.6 [1.9 to 3.6] | 2.5 [1.5 to 3.4] | 5.2 [1.2 to 12.6] | 4.3 [3.5 to 5.1] | 2.9 [2.9 to 2.9] | 2.8 [2.6 to 3.0] | 6.8 [2.7 to 14.3]
  135 min | 4.0 [3.0 to 4.9] | 2.2 [2.1 to 2.3] | 2.6 [2.3 to 2.9] | 5.0 [1.2 to 12.1] | 3.8 [2.9 to 4.7] | 2.7 [2.7 to 2.7] | 2.6 [2.6 to 2.7] | 7.4 [2.7 to 16.5]
  150 min | 2.9 [2.9 to 3.0] | 7.8 [2.3 to 18.4] | 2.0 [1.4 to 2.6] | 5.0 [1.2 to 12.2] | 3.7 [2.9 to 4.4] | 2.6 [2.6 to 2.6] | 2.6 [2.5 to 2.7] | 7.0 [2.8 to 13.4]
  165 min | 3.1 [2.7 to 3.4] | 2.6 [2.1 to 3.7] | 2.6 [2.4 to 2.8] | 5.0 [1.1 to 12.0] | 4.6 [4.1 to 5.1] | 2.6 [2.6 to 2.6] | 2.6 [2.5 to 2.6] | 3.4 [2.6 to 4.1]
  180 min | 3.1 [2.9 to 3.4] | 2.1 [1.8 to 2.4] | 2.1 [1.4 to 2.7] | 4.8 [1.2 to 11.5] | 3.3 [2.7 to 3.9] | 2.6 [2.6 to 2.6] | 2.6 [2.5 to 2.6] | 3.2 [2.7 to 3.5]
  195 min | 3.8 [3.0 to 4.6] | 4.0 [1.8 to 8.3] | 2.5 [1.5 to 3.4] | 5.2 [1.1 to 12.8] | 3.8 [3.1 to 4.4] | 2.6 [2.6 to 2.6] | 2.6 [2.5 to 2.8] | 3.4 [2.7 to 4.5]
  210 min | 3.6 [3.1 to 4.2] | 4.0 [1.8 to 7.0] | 2.2 [1.9 to 2.4] | 4.8 [1.2 to 11.7] | 3.9 [2.9 to 4.9] | 2.8 [2.8 to 2.8] | 2.6 [2.5 to 2.7] | 6.3 [2.7 to 8.6]
  225 min | 3.4 [3.1 to 3.6] | 4.3 [1.7 to 9.1] | 1.9 [1.5 to 2.3] | 4.9 [1.1 to 12.0] | 3.1 [2.9 to 3.3] | 2.4 [2.4 to 2.4] | 2.6 [2.5 to 2.7] | 3.3 [2.7 to 4.0]
  240 min | 3.2 [3.0 to 3.5] | 3.9 [1.7 to 8.0] | 2.9 [1.4 to 4.3] | 7.4 [1.2 to 10.9] | 3.4 [2.6 to 4.2] | 2.6 [2.6 to 2.6] | 2.5 [2.5 to 2.6] | 5.3 [2.6 to 9.3]
  255 min | 3.1 [2.6 to 3.6] | 4.0 [1.6 to 8.7] | 8.5 [1.3 to 15.6] | 4.8 [1.1 to 11.8] | 3.8 [2.7 to 4.8] | 2.5 [2.5 to 2.5] | 2.9 [2.7 to 3.0] | 4.9 [2.7 to 9.1]
  270 min | 3.3 [3.2 to 3.4] | 4.4 [1.7 to 9.4] | 8.8 [1.9 to 15.6] | 5.0 [1.5 to 11.9] | 3.5 [2.5 to 4.4] | 2.7 [2.7 to 2.7] | 2.5 [2.4 to 2.6] | 4.8 [2.6 to 8.8]
  285 min | 2.9 [2.8 to 3.0] | 4.9 [2.0 to 10.7] | 1.9 [1.4 to 2.5] | 4.4 [1.2 to 10.4] | 2.8 [2.5 to 3.1] | 2.5 [2.5 to 2.5] | 2.6 [2.6 to 2.6] | 4.3 [2.7 to 7.6]

2. Secondary Outcome: Number of Attempts Needed for Successful Subcutaneous Catheter/Needle Placement
Time Frame: end of catheter/needle placement
Population: Per Protocol (two subjects excluded due to technical error in in-line fluid pressure measurements)
Measure: Number; unit: Subjects
Arm/Group | 24 ga Catheter, Dose Flush, Single-step Rate Scheme | 24 ga Catheter, No Dose Flush, Single-step Rate Scheme | 24 ga Catheter, Dose Flush, Up-titrated Rate Scheme | 24 ga Catheter, No Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, Dose Flush, Single-step Rate Scheme | 25 ga Needle, No Dose Flush, Single-step Rate Scheme | 25 ga Needle, Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, No Dose Flush, Up-titrated Rate Scheme
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 1 | 2 | 3
Subjects
  1 attempt | 2 | 3 | 2 | 2 | 2 | 1 | 2 | 3
  2 attempts | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

3. Secondary Outcome: Cumulative Fluid Volume Delivered
Time Frame: as for outcome 1
Population: Per Protocol (two subjects excluded due to technical errors in fluid pressure measurement)
Measure: Mean (Full Range); unit: mL
Arm/Group | 24 ga Catheter, Dose Flush, Single-step Rate Scheme | 24 ga Catheter, No Dose Flush, Single-step Rate Scheme | 24 ga Catheter, Dose Flush, Up-titrated Rate Scheme | 24 ga Catheter, No Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, Dose Flush, Single-step Rate Scheme | 25 ga Needle, No Dose Flush, Single-step Rate Scheme | 25 ga Needle, Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, No Dose Flush, Up-titrated Rate Scheme
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 1 | 2 | 3
mL
  5 min | 20.8 [20.7 to 20.8] | 21.4 [20.6 to 22.2] | 4.2 [4.2 to 4.2] | 3.8 [3.1 to 4.2] | 21.1 [21.1 to 21.1] | 20.7 [20.7 to 20.7] | 4.1 [4.1 to 4.1] | 4.1 [4.1 to 4.2]
  10 min | 41.2 [41.2 to 41.2] | 41.3 [39.6 to 42.9] | 11.7 [11.4 to 11.9] | 11.5 [10.4 to 12.3] | 42.0 [41.9 to 42.1] | 41.2 [41.2 to 41.2] | 12.1 [12.0 to 12.1] | 11.9 [11.8 to 12.1]
  60 min | 250 [249 to 250] | 249 [248 to 250] | 249 [248 to 249] | 240 [228 to 247] | 249 [247 to 250] | 249 [249 to 249] | 248 [247 to 248] | 246 [243 to 248]
  120 min | 448 [447 to 449] | 450 [448 to 452] | 449 [447 to 451] | 447 [447 to 448] | 449 [448 to 450] | 447 [447 to 447] | 448 [446 to 449] | 446 [441 to 448]
  180 min | 649 [647 to 650] | 650 [648 to 652] | 649 [647 to 651] | 647 [647 to 648] | 649 [648 to 650] | 647 [647 to 647] | 650 [649 to 650] | 646 [641 to 648]
  240 min | 848 [847 to 849] | 850 [848 to 853] | 849 [847 to 851] | 848 [847 to 849] | 849 [848 to 850] | 847 [847 to 847] | 847 [845 to 848] | 846 [841 to 848]
  285 min | 998 [995 to 1000] | 1000 [998 to 1002] | 999 [997 to 1000] | 997 [997 to 998] | 999 [998 to 1000] | 997 [997 to 997] | 997 [997 to 997] | 996 [991 to 998]

4. Secondary Outcome: Technical Challenges Encountered During Fluid Infusion
Description: Observed challenges, including catheter kinking, catheter/needle dislodgement/pull-out, infusion pump alarm, other technical problems
Time Frame: at any occurence of a defined challenge or at end of infusion if no challenges occurred
Population: Per Protocol (two subjects excluded due to technical error in in-line fluid pressure measurement)
Measure: Number; unit: participants
Arm/Group | 24 ga Catheter, Dose Flush, Single-step Rate Scheme | 24 ga Catheter, No Dose Flush, Single-step Rate Scheme | 24 ga Catheter, Dose Flush, Up-titrated Rate Scheme | 24 ga Catheter, No Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, Dose Flush, Single-step Rate Scheme | 25 ga Needle, No Dose Flush, Single-step Rate Scheme | 25 ga Needle, Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, No Dose Flush, Up-titrated Rate Scheme
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 1 | 2 | 3
participants
  Any Technical Challenge | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Catheter Kinking | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Occlusion Alarm | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Intervention Needed to Secure/Maintain Infusion | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | 24 ga Catheter, Dose Flush, Single-step Rate Scheme | 24 ga Catheter, No Dose Flush, Single-step Rate Scheme | 24 ga Catheter, Dose Flush, Up-titrated Rate Scheme | 24 ga Catheter, No Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, Dose Flush, Single-step Rate Scheme | 25 ga Needle, No Dose Flush, Single-step Rate Scheme | 25 ga Needle, Dose Flush, Up-titrated Rate Scheme | 25 ga Needle, No Dose Flush, Up-titrated Rate Scheme
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/3 | 0/3 | 0/2 | 0/2 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 3/3 | 3/3 | 2/2 | 2/2 | 2/2 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 24 ga Catheter, Dose Flush, Single-step Rate Scheme (N=2) | 24 ga Catheter, No Dose Flush, Single-step Rate Scheme (N=3) | 24 ga Catheter, Dose Flush, Up-titrated Rate Scheme (N=3) | 24 ga Catheter, No Dose Flush, Up-titrated Rate Scheme (N=3) | 25 ga Needle, Dose Flush, Single-step Rate Scheme (N=2) | 25 ga Needle, No Dose Flush, Single-step Rate Scheme (N=2) | 25 ga Needle, Dose Flush, Up-titrated Rate Scheme (N=2) | 25 ga Needle, No Dose Flush, Up-titrated Rate Scheme (N=3)
Infusion site erythema (General disorders) | 2 | 3 | 3 | 3 | 2 | 2 | 2 | 2/2
Infusion site oedema (General disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 1
Infusion site pain (General disorders) | 2 | 3 | 2 | 2 | 2 | 0 | 2 | 2
Infusion site pruritus (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Infusion site rash (General disorders) | 1 | 3 | 1 | 2 | 1 | 0 | 1 | 1
Infusion site swelling (General disorders) | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to small numbers of subjects in each treatment arm, no conclusions can be drawn on the influence of any of the individual potential pressure-affecting factors or the combinations of these factors on in-line fluid pressure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For this study, Baxter requires a review of any planned PI results communications (eg, for confidential information) up to 30 days prior to submission or communication. Baxter may request an additional delay of up to 60 days (eg, to allow for intellectual property protection).